CLINICAL TRIAL: NCT03646786
Title: Prospective Pilot Study of Multi-actor Tolerance Evaluation Using the VIRARE Device (VIrtual Reality Assisted Rehabilitation) in Visually Impaired Patients
Acronym: VIRARE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IDIL/2016/LJ-01
Record Dates: First submitted 2018-08-23; First posted 2018-08-24 (Actual); Last update posted 2022-09-28 (Actual); Status verified 2022-09

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- visually impaired patients (Experimental)
  Interventions: Device: Virtual reality tests

INTERVENTIONS:
Device: Virtual reality tests — The patient will complete 3 self-questionnaires and pass 3 exploratory tests of virtual reality:
  1. 10 minutes sitting test: detection of 5 targets in a 360 ° field of vision
  2. 10-minute stand-up motionless test: detection of 5 targets in a 360 ° field of view and placing ingredients of a recipe
  3. Standing 10-minute test: the patient moves to the site of his mission, detection of 5 targets in a 360 ° field of vision and preparing a recipe

SUMMARY:
Our study aims to validate the relevance of a virtual reality tool (VIRARE: VIrtual REality Assisted Rehabilitation) in the assessment and rehabilitation of visually impaired subjects.

ELIGIBILITY:
Inclusion Criteria:

* The patient signed the consent form
* The patient is affiliated to a health insurance programme
* The patient presents ophthalmological or neurological pathologies with impact on visual function (retinopathy pigmentosa, macular dystrophy, glaucoma, age-related macular degeneration, cerebrovascular accident ...).
* The patient is visually impaired (visual acuity less than 3/10 of both eyes or concentric narrowing of the Goldmann binocular visual field or homonymous hemianopia) of category I, II, III or IV of the WHO classification.

Exclusion Criteria:

* The patient is participating in another study
* The patient is in an exclusion period determined by another study
* The patient is under safeguard of justice.
* The patient is under judicial protection.
* It is not possible to give the patient (or his/her trusted-person) informed information.
* The patient is pregnant or breastfeeding.
* The patient has a sensory or cognitive disability with a given scale (MMS < 24)
* The patient has difficulty moving including major locomotor difficulties.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2020-12-11 (Actual); Primary Completion 2021-11-12 (Actual); Study Completion 2022-03-11 (Actual)

PRIMARY OUTCOMES:
dizziness felt by the patient | Day 0
  Yes/no
Nausea felt by the patient | Day 0
  Yes/no
headache felt by the patient | Day 0
  Yes/no
dazzle felt by the patient | Day 0
  Yes/no
watering of the patient | Day 0
  Yes/no
eye burns felt by the patient | Day 0
  Yes/no
Pain due to the mobilization of the eyeballs felt by the patient | Day 0
  Yes/no
Extraocular pain felt by the patient | Day 0
  Yes/no
diplopia | Day 0
  Yes/no
amaurosis | Day 0
  Yes/no
Fear | Day 0
  Yes/no
conformity of the session according to the patient point of view | Day 0
  Yes/no
unpleasantness of the session from the patient point of view | Day 0
  Yes/no
Difficulty of the session according to the patient point of view | Day 0
  Yes/no
Willingness to continue the following tests according to the patient point of view | Day 0
  Yes/no
Cervical pain felt by the patient | Day 0
  Yes/no
oculomotricity of the patient according to the therapist | Day 0
  Rank: 0-missing, 1-insufficient, 2-medium, 3-suitable
head movements of the patient according to the therapist | Day 0
  Rank: 0-missing, 1-insufficient, 2-medium, 3-suitable
body movements of the patient according to the therapist | Day 0
  Rank: 0-missing, 1-insufficient, 2-medium, 3-suitable
target tracking by the patient according to the therapist | Day 0
  0 = 0 target detected
  1. 1 or 2 targets detected
  2. 3 or 4 targets detected
  3. 5 targets detected
Time lapse to find targets | Day 0
  minutes
The patient asked for a pause during the test | Day 0
  Yes/no
The patient asked to permanently stop the tests | Day 0
  Yes/no
The patient went to the right place during the 3rd test | Day 0
  Yes/no
The patient has correctly performed the requested task | Day 0
  Yes/no

CONTACTS AND LOCATIONS:
Overall Officials: Luc JEANJEAN, Principal Investigator — Nîmes University Hospital
Locations (1):
- Nimes University Hospital, Nîmes, France